CLINICAL TRIAL: NCT05387343
Title: COVID Vaccine Immunity in Kidney Transplant Recipients
Status: Withdrawn | Type: Observational
Why Stopped: funding lost
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: ViraCor Laboratories (Industry)
Responsible Party: Principal Investigator, Graham C. Towns, Associate Professor, University of Alabama at Birmingham
Other Study IDs: GCT2022.001
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: End Stage Renal Disease; Kidney Transplant; Complications
Keywords: COVID-19; kidney; kidney transplant; end stage renal disease; mRNA vaccine
MeSH Terms: conditions — Kidney Failure, Chronic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples will be collected for spike protein antibodies and t cell assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronavirus (COVID-19) SARS-CoV-2 inSIGHT™ T Cell Immunity Test — Boosters will be given after month 3 after transplant, and the 2nd booster will be given 3 months after the first.
  Other Names: mRNA COVID vaccine

SUMMARY:
50 end-stage renal disease (ESRD) patients whom have had at least 2 doses of messenger ribonucleic acid (mRNA) vaccine, and undergoing transplantation at the University of Alabama at Birmingham (UAB) will be enrolled. The third mRNA vaccine will be given 3 months post transplant, and the 4th mRNA vaccine will be given 3 months following this. Blood samples will be collected and shipped to Viracor on day of transplant, and at months 1, 3, 4, 6, and 12 for spike protein and t cell assay.

DETAILED DESCRIPTION:
50 ESRD patients on peritoneal dialysis or hemodialysis or not on immunosuppression, no prior transplant, no known history of COVID infection, whom have had at least 2 doses of mRNA vaccine, and undergoing transplantation at UAB will be enrolled, after signing the informed consent. The third mRNA vaccine will be given 3 months post transplant, and the 4th mRNA vaccine will be given 3 months following this. Blood samples will be collected and shipped to Viracor on day of transplant, and at months 1, 3, 4, 6, and 12 for spike protein and t cell assay.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Renal Disease patients on peritoneal dialysis or hemodialysis or not on immunosuppression
* no prior transplant
* no known history of COVID infection
* had at least 2 doses of mRNA COVID vaccine
* undergoing transplantation at the University of Alabama at Birmingham
* multi-organ transplant allowed

Exclusion Criteria:

* active COVID infection
* participant is not vaccinated against COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients planning on having a renal transplant at the University of Alabama at Birmingham
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
COVID spike protein Immunoglobulin G (IgG) and Tcell assay | pre-transplant
  transplant patient response to vaccine compared to response of patients not on immunosuppression
COVID spike protein IgG and Tcell assay | month 1
  transplant patient response to vaccine compared to response of patients not on immunosuppression
COVID spike protein IgG and Tcell assay | month 3
  transplant patient response to vaccine compared to response of patients not on immunosuppression
COVID spike protein IgG and Tcell assay | month 4
  transplant patient response to vaccine compared to response of patients not on immunosuppression
COVID spike protein IgG and Tcell assay | month 6
  transplant patient response to vaccine compared to response of patients not on immunosuppression
COVID spike protein IgG and Tcell assay | month 12
  transplant patient response to vaccine compared to response of patients not on immunosuppression

CONTACTS AND LOCATIONS:
Overall Officials: Graham C Towns, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No